CLINICAL TRIAL: NCT00969410
Title: A Pharmacodynamic Study of AV-299 (Formerly SCH 900105) in Subjects With Advanced Solid Tumors Who Have Liver Metastases (P05670)
Brief Title: A Pharmacodynamic Study of AV-299 (Formerly SCH 900105) in Subjects With Advanced Solid Tumors Who Have Liver Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05670
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Malignant Solid Tumour; Liver Metastases
Keywords: Neoplasms; Neoplasm metastasis; Liver neoplasms; Neoplastic processes; Pathologic processes; Digestive system neoplasms; Neoplasms by site; Digestive system diseases; Liver diseases
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Liver Neoplasms; Neoplastic Processes; Pathologic Processes; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Liver Diseases | interventions — ficlatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AV-299 administered IV (monotherapy) (Experimental): Subjects will be enrolled sequentially and treated with AV-299 (formerly SCH 900105) in dose escalating cohorts. Accrual to the next cohort will occur only if <= 1 out of 6 subjects experiences a dose-limiting toxicity (DLT) during the first 2 cycles. If >= 2 subjects in the same dose cohort experience a DLT during the first 2 cycles, dose-escalation will be terminated.
  Interventions: Biological: AV-299

INTERVENTIONS:
Biological: AV-299 — AV-299 will be given as an intravenous infusion in dose-escalating doses of 2, 10, and 20 mg/kg once every 2 weeks.
  Other Names: Ficlatuzumab, Formerly SCH900105

SUMMARY:
A pharmacodynamic study to evaluate the effect of AV-299 on exploratory pharmacodynamic markers in subjects with advanced solid tumors who have liver metastases.

To evaluate safety and tolerability of AV-299 administered IV in subjects with advanced solid tumors who have liver metastases.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give written informed consent and be able to adhere to dose and visit schedules.
* Diagnosis of an advanced colorectal, breast, gastric/esophageal or pancreatic cancer with liver metastases that are amenable to biopsy.
* Histological or cytological evidence of malignancy.
* Advanced metastatic colorectal, breast, gastric/esophageal or pancreatic cancer that has recurred or progressed following standard therapy or failed standard therapy; or for which no standard therapy currently exists, or for which subject is not a candidate for, or is unwilling to undergo standard therapy.

Note: Additional tumor histologies may be eligible based on available HGF/c-Met pathway data and approval by the Sponsor.

* Disease that is currently not amenable to curative surgical intervention.
* Male or female and ≥ 18 years of age.
* ECOG performance status of 0-1.
* Measurable p-Met by immunohistochemistry in archived or otherwise available tumor sample.
* Female subjects of childbearing potential must have negative pregnancy test within 5 days prior to first dose of study drug.
* Female subjects of childbearing potential and male subjects whose sexual partners are of childbearing potential must agree to abstain from sexual intercourse or to use an effective method of contraception during the study and for 60 days after the last dose of AV-299 (formerly SCH 900105). Examples of effective methods of contraception include oral contraceptives or double barrier methods such as condom plus spermicide or condom plus diaphragm.
* Adequate hematologic function as evidenced by Hg ≥ 9g/dL, WBC ≥ 3000 per mm3, ANC ≥ 1500 per mm3 and platelet count ≥ 100,000 per mm3.
* Adequate hepatic function as evidenced by a serum bilirubin level ≤ 1.5 × ULN (except with known Gilbert's Syndrome) and with serum AST/ALT levels ≤ 5 × ULN.
* Adequate renal function as evidenced by a serum creatinine level ≤ 1.5 × ULN or a calculated creatinine clearance > 60 mL/min.
* Adequate coagulation function as evidenced by PTT ≤ 1.5 × ULN and INR ≤ 1.5 × ULN.
* Recovery from the effects of any prior surgery, radiotherapy, or systemic antineoplastic therapy.
* Subjects with abnormal liver function tests (LFTs) who have not been screened for Hepatitis B or C within the past 6 months prior to study enrollment, will need to be screened for Hepatitis B and C and can only be enrolled if the screening is negative.

Exclusion Criteria:

* Women who are breast-feeding, pregnant, or intend to become pregnant.
* Hematologic malignancies.
* Any of the following within 6 months prior to administration of study drug:
* Myocardial infarction (MI), severe/unstable angina pectoris, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack or seizure disorder.
* Serious/symptomatic active infection, or infection requiring antibiotics, within 14 days prior to first dose of study drug.
* Persistent, unresolved CTCAE v3.0 Grade 2 or higher drug-related toxicity (except alopecia, erectile dysfunction, hot flashes, decreased libido, and Grade 2 sensory peripheral neuropathy) associated with previous treatment.
* Inadequate recovery from any prior surgical procedure or major surgical procedure performed within 4 weeks prior to administration of first dose of study drug.
* Any other medical or psychiatric condition that, in the opinion of the investigator, might interfere with the subject's participation in the trial or interfere with the interpretation of trial results.
* Known Human Immunodeficiency Virus (HIV) infection or a known HIV-related malignancy.
* Known active hepatitis B or C.
* Known hypersensitivity to any of the components of SCH 900105.
* Known bleeding diathesis.
* Radiotherapy within 3 weeks prior to first study drug administration.
* Inability to comply with the protocol requirements, including inability to undergo liver biopsies.
* Participation in any other clinical trials involving therapeutic agents.
* Any medications prohibited in the study.
* Active alcohol or illicit drug abuse.
* Stem cell/bone marrow transplant within 6 months of first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of AV-299 (formerly SCH 900105) on exploratory pharmacodynamic markers in subjects with advanced solid tumors who have liver metastases | Screening Cycle 1: Day 1, Day 3-4: Cycle 2: Day 1 Cycle 3: Day 8-14
  Peripheral blood analysis, liver tissue analysis, and PET
To evaluate safety and tolerability of AV-299 (formerly SCH 900105) administered IV in subjects with advanced solid tumors who have liver metastases | DLTs assessed during first 4 weeks of treatment.
  Dose-limiting toxicities.

SECONDARY OUTCOMES:
To evaluate the PK of AV-299 (formerly SCH 900105) in subjects with advanced solid tumors who have liver metastases | Cycle 1: Day 1, Day 3-4 Cycle 2: Day 1 Cycle 3: Day 1, Day 8-14
To study the preliminary antineoplastic activity of AV-299 (formerly SCH 900105) in subjects with advanced solid tumors who have liver metastases | Subjects will undergo disease assessment at screening (within 4 weeks prior to first dose of study drug), the Cycle 3 Day 8-14 visit, and approximately every 6 weeks thereafter.
To investigate the effect of AV-299 (formerly SCH 900105) on gene expression patterns in peripheral blood mononuclear cells and liver biopsies in subjects with advanced solid tumors who have liver metastases | Cycle 1: Day 1, Day 3-4 Cycle 3: Day 8-14:

CONTACTS AND LOCATIONS:
Overall Officials: Shefali Agarwal, MD, Study Director — AVEO Pharmaceuticals, Inc.
Locations (1):
- Investigational Site 1, Barcelona, Spain